CLINICAL TRIAL: NCT01475383
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study Of The Safety And Efficacy Of PF-03654746 In Adults With Tourette's Syndrome
Brief Title: Study Evaluating The Safety And Efficacy Of PF-03654746 In Adult Subjects With Tourette's Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A8801035
Record Dates: First submitted 2011-10-25; First posted 2011-11-21 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Tourette's Syndrome
Keywords: Tourette's Syndrome in adults; Safety and Efficacy; Randomized; Placebo Control; Cross-over
MeSH Terms: conditions — Tourette Syndrome | interventions — N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-03654746 (Active Comparator): Subjects are randomized to either active drug or placebo in Period 1; in Period 2 the sequence is reversed.
  Interventions: Drug: PF-03654746; Drug: Placebo
- Placebo (Placebo Comparator): Subjects are randomized to either active drug or placebo in Period 1; in Period 2 the sequence is reversed.
  Interventions: Drug: Placebo; Drug: PF-03654746

INTERVENTIONS:
Drug: PF-03654746 — 20-day dose titration phase: all dosages in capsules starting at 0.25 mg qd x 5 d, then 0.5 mg qd x 5 d, then 1.0 mg qd x 5 d, then 2.0 mg qd x 5 d. If a subject has intolerable, severe, or serious AEs after taking 2 mg qd for 1 to 5 days of dosing, the dose will be decreased by the investigator to 1 mg qd. If, in the investigator's opinion, the subject is determined to be unlikely to tolerate continued dosing at a dose of 1 mg qd, the subject should be discontinued from the study. Subjects remaining in the study will proceed to the 3-week Stable Dosing Phase; doses will be 2 mg daily x 21 days or 1 mg daily x 21 days.
  Arms: PF-03654746
Drug: Placebo — once daily dosing of placebo capsules following the dosing scheme described in 1.1.
  Arms: PF-03654746
Drug: Placebo — once daily dosing of placebo capsules following the dosing scheme described in 1.1
  Arms: Placebo
Drug: PF-03654746 — 20-day dose titration phase: all dosages in capsules starting at 0.25 mg qd x 5 d, then 0.5 mg qd x 5 d, then 1.0 mg qd x 5 d, then 2.0 mg qd x 5 d. If a subject has intolerable, severe, or serious AEs after taking 2 mg qd for 1 to 5 days of dosing, the dose will be decreased by the investigator to 1 mg qd. If, in the investigator's opinion, the subject is determined to be unlikely to tolerate continued dosing at a dose of 1 mg qd, the subject should be discontinued from the study. Subjects remaining in the study will proceed to the 3-week Stable Dosing Phase; doses will be 2 mg daily x 21 days or 1 mg daily x 21 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an investigational compound designated PF-03654746 compared to placebo in the treatment of adults with Tourette's Syndrome. The study will also explore the pharmacokinetics of PF-03654746 in adults with Tourette's Syndrome.

DETAILED DESCRIPTION:
The study was terminated 11-Apr-2012 due to an internal reassessment of priorities by the sponsor. The decision to terminate was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Tourette's Syndrome in English-speaking male or female adults 18 to 55 years of age who are in generally good health.
* Free of medications to treat tics for at least 6 weeks prior to randomization.
* Females of childbearing potential must use medically acceptable birth control for the duration of the study and for 28 days after study participation.

Exclusion Criteria:

* Tic treatment including protocol-specified drugs, training in tic-suppressing behavioral techniques, habit reversal training or use of Onabotulinum toxin A injection.
* History or neurologic evidence of a secondary tic disorder, psychosis, bipolar disorder, tardive dyskinesia, untreated or unstable DSM-IV Axis I disorder requiring treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in Total Tic Score (Yale Global Tic Severity Scale) from baseline (D0) to end of the 3 wk stable dosing phase (D41)(primary). Average of the 2 assessments of Total Tic Score in 3 wk stable dosing phase is secondary. Score 0-50 (50 = severe) | Period 1: Days 0, 10, 20, 34, 41; Period 2: Days 0, 10, 20, 34, 41

SECONDARY OUTCOMES:
Change in Tic Symptom Self Report from baseline to end of 3-wk stable dosing phase (primary); average of 2 assessments of TSSR during 3-wk stable dosing phase is 2ndary. Each symptom is scored 0-3; higher score is worse. | Period 1: Days 0, 10, 20, 34, 41; Period 2: Days 0, 10, 20, 34, 41
Change in Premonitory Urge for Tic Scale from baseline to end of 3-wk stable dosing phase (primary); average of 2 assessments of PUTS during 3-wk stable dosing phase is 2ndary. Score 9-36; higher score is worse. | Period 1: Days 0, 10, 20, 34, 41; Period 2: Days 0, 10, 20, 34, 41
Change in Clinical Global Impression of Severity from baseline to end of 3-wk stable dosing phase. Score 1-7; higher scores indicate more severity. | Period 1, Days 0, 41; Period 2: Days 0, 41
Change in Clinical Global Impression of Improvement from baseline to end of 3-wk stable dosing phase (primary); average of 2 assessments during 3-wk stable dosing phase is 2ndary. Score 1-7; higher score is worse. | Period 1: Days 10, 20, 34, 41; Period 2: Days 10, 20, 34, 41
Change in Conners' Continuous Performance Test II from baseline to end of 3-wk stable dosing phase. Calculated T-scores (under 40 to 65 and over); higher score is worse. | Period 1: Days 0, 20, 41; Period 2: Days 0, 20, 41
Change in Medical Outcomes Study--Sleep Scale from baseline to end of 3-wk stable dosing phase. Score 0-100; a higher score reflect greater amount of quality implied by subscale name. | Period 1: Days 0, 10, 20, 34, 41; Period 2: Days 0, 10, 20, 34, 41
Change in Columbia Suicide Severity Rating Scale from baseline to end of 3-wk stable dosing phase. | Screening; Period 1: Days 0, 10, 20, 34, 41; Period 2: Days 0, 10, 20, 34, 41
Suicide Behaviors Questionnaire-Revised. Total score greater than 8 require assessment by clinician or mental health professional skilled in evaluation of suicidality. | Up to 21 days prior to Baseline (Day 0)
Change in Yale-Brown Obsessive-Compulsive Scale from baseline to end of 3-wk stable dosing phase. Items 1-10 have score range of 0-40; higher score is worse. | Period 1: Days 0, 41; Period 2: Days 0, 41

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Manhasset, New York, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8801035&StudyName=Study%20Evaluating%20The%20Safety%20And%20Efficacy%20Of%20PF-03654746%20In%20Adult%20Subjects%20With%20Tourette%27s%20Syndrome